CLINICAL TRIAL: NCT00626223
Title: 5-methyltetrahydrofolate Survival and Inflammation in ESRD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: University of Bologna (Other)
Responsible Party: Professor Sergio Stefoni, Nephrology Dialysis and Renal Transplantation Unit, S.Orsola University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FCRB 2007/0234; ndtso 00025/2007
Record Dates: First submitted 2008-02-04; First posted 2008-02-29 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Mortality; Hyperhomocysteinemia; Inflammation
Keywords: ESRD patients; C-reactive protein; homocysteine; 5-MTHF; survival; Hemodialysis patients
MeSH Terms: conditions — Hyperhomocysteinemia; Inflammation | interventions — 5-methyltetrahydrofolate; Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): patients treated with intravenous 5-MTHF (Prefolic®, Knoll, Milan, Italy) 50 mg at the end of each hemodialysis session; The group will receive supplementation with vitamin B6 300 mg (Benadon®, Roche, Milan, Italy) and vitamin B12 1000 mcg (Dobetin®, A.C.R.A.F, Rome, Italy) administered by intravenous injection at the end of the hemodialysis session three times per week
  Interventions: Drug: 5-MTHF (5-methyltetrahydrofolate)
- B (Active Comparator): treated with 5 mg per day of oral folic acid (Folina® Schwarz Pharma, Milan, Italy).
  The group will receive supplementation with vitamin B6 300 mg (Benadon®, Roche, Milan, Italy) and vitamin B12 1000 mcg (Dobetin®, A.C.R.A.F, Rome, Italy) administered by intravenous injection at the end of the hemodialysis session three times per week
  Interventions: Drug: folic acid

INTERVENTIONS:
Drug: 5-MTHF (5-methyltetrahydrofolate) — 50 mg intravenous at the end of each hemodialysis session
  Arms: A
Drug: folic acid — 5 mg per day of oral folic acid
  Arms: B

SUMMARY:
A randomized prospective study was done to determine whether i.v. 5-methyltetrahydrofolate vs oral folate improved survival in ESRD patients. Homocysteine, CRP, Lp(a), albumin, folates, vitamin B6 and B12 were checked. The 5-MTHF treated group was associated with lowered C reactive protein and higher survival than the folate treated group.

DETAILED DESCRIPTION:
BACKGROUND Hemodialysis patients show a 20-fold increase in CVD mortality in comparison to the general population.

Although hyperhomocysteinemia has been implicated as an important independent risk factor in both the general population2, as well as for ESRD patients, several studies have questioned the benefit of lowering homocysteine in ESRD patients. Paradoxically, two recent studies showed that patients with very low homocysteine plasma levels had worse outcomes including a higher incidence of hospitalization and mortality. This raises the question as to whether elevated homocysteine in uremic patients is consequential rather than causal in the role of cardiovascular complications.

Despite this uncertainty, many ESRD and pre-ESRD patients receive treatment to lower homocysteine. Elevated homocysteine is frequently reported for ESRD patients with a prevalence ranging from 85 to 100%.

There are two basic strategies that can be used to lower homocysteine. Both attempt to increase levels of biologically active folate which is essential in the remethylation pathway of homocysteine metabolism via its active metabolite 5-methyltetrahydrofolate (5-MTHF), thus lowering homocysteine efflux from tissues into the plasma compartment.

The first, and most common approach, is by oral administration of folic acid. Folic acid is not biologically active, however it is more stable than folate, and is often used in tablets and food fortification. The second approach is to supplement 5-MTHF, the natural circulating form of folate. In addition to folate, both vitamin B6 and vitamin B12 are necessary co-factors in homocysteine metabolism. ESRD patients are often resistant to homocysteine lowering by administration of both folic acid and 5-MTHF.

Although supplementation with folic acid, B6 and B12 usually decreases homocysteine in patients with vascular disease, it often remains elevated in ESRD patients despite supplementation of folic acid, B6 and B12. Several studies have reported only moderate effects, even with very high doses of folic acid (up to 15 mg/daily).

AIM OF THE STUDY The aim of this study is to investigate whether supplementation with 5MTHF vs. folic acid treatment affects patient survival. Homocysteine blood levels and MTHFR genetic polymorphisms will also be evaluated to determine if they can be considered as independent cardiovascular risk factors.

STUDY DESIGN Single center, randomised, prospective study. Two groups of stable ESRD patients treated with intravenous 5-MTHF or with 5 mg per day of oral folic acid.

Patient selection Period of selection : 4 years Start selection : 1 January 1998 End selection: 30 June 2001 Follow-up: 55 months.

STATISTICAL ANALYSIS Statistical analysis will be performed by the Statistical Package for the Social Sciences (SPSS).

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patients with age > 18 years on regular bicarbonate hemodialysis or hemodiafiltration treatment three times a week
* Clinical stability at least three months before the study started
* Cardiovascular disease assessment as presence/absence of hypertension, ischemic cardiac disease, cerebral and peripheral vascular disease, diabetes.

  * We will investigate coronary artery disease by determination of at least one of the following parameters:

    * previous documentation of acute myocardial infarction (laboratory or ECG modifications);
    * symptomatic CVD events in the clinical history confirmed by a positive treadmill test;
    * coronary artery stenosis more than 50% in one of the three major coronary vessels documented by an angiographic study. All patients with coronary artery disease will be examined by a treadmill test (thallium scan) or coronary angiographic exam before entering the study.
  * We will investigate cerebrovascular disease by one of the following criteria:

    * a previous ictus (ongoing clinical evidence of neurological deficit in the three months before the study beginning, confirmed by a TC scan, a nuclear magnetic resonance or a physician's record of clinical history);
    * carotid vessels stenosis more than 50% documented by a Doppler exam.
  * Peripheral vascular disease will be assessed by the evidence of claudication intermittence, previous vascular surgical procedure (including amputation for ischemic limb or by angiographic/Doppler documentation of atherosclerotic plaques in abdominal, iliac and femoral vessels). The vascular surgical procedure will be carried out at least three months before the study started.

Exclusion Criteria:

* Diagnosis of one of the following clinical conditions in the last three months:

  * acute infection
  * vascular access thrombosis
  * ictus cerebri
  * myocardial infarction
  * hemorrhage
  * recent relevant surgery
* Malignancy
* Participation in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 1998-01; Primary Completion 2001-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
survival | 55 months

SECONDARY OUTCOMES:
Risk factors for cardiovascular disease in ESRD patients | 55 months
Homocysteine levels after 6, 12, 24 and 55 months | 55 months
CRP levels after 6, 12, 24 and 55 months | 55 months
Gene polymorphisms analysis on C677T and A1298C loci and differences in polymorphisms distribution in both groups | basal
Differences at baseline between the groups concerning age, dialysis age, CRP, albumin, haemoglobin, Lp(a), homocysteine, folate, B6 and B12 baseline levels | basal

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Stefoni, Professor, Study Chair — Nephrology Dialysis and Renal Trasnplantation Unit S.Orsola University Hospital Bologna Italy
Locations (1):
- Nephrology Dialysis and Renal Transplantation Unit, S.Orsola University Hospital, Bologna, Italy

REFERENCES:
- [Background] Cheung AK, Sarnak MJ, Yan G, Berkoben M, Heyka R, Kaufman A, Lewis J, Rocco M, Toto R, Windus D, Ornt D, Levey AS; HEMO Study Group. Cardiac diseases in maintenance hemodialysis patients: results of the HEMO Study. Kidney Int. 2004 Jun;65(6):2380-9. doi: 10.1111/j.1523-1755.2004.00657.x. PMID 15149351
- [Background] Nygard O, Vollset SE, Refsum H, Stensvold I, Tverdal A, Nordrehaug JE, Ueland M, Kvale G. Total plasma homocysteine and cardiovascular risk profile. The Hordaland Homocysteine Study. JAMA. 1995 Nov 15;274(19):1526-33. doi: 10.1001/jama.1995.03530190040032. PMID 7474221
- [Background] Buccianti G, Baragetti I, Bamonti F, Furiani S, Dorighet V, Patrosso C. Plasma homocysteine levels and cardiovascular mortality in patients with end-stage renal disease. J Nephrol. 2004 May-Jun;17(3):405-10. PMID 15365961
- [Background] Mallamaci F, Bonanno G, Seminara G, Rapisarda F, Fatuzzo P, Candela V, Scudo P, Spoto B, Testa A, Tripepi G, Tech S, Zoccali C. Hyperhomocysteinemia and arteriovenous fistula thrombosis in hemodialysis patients. Am J Kidney Dis. 2005 Apr;45(4):702-7. doi: 10.1053/j.ajkd.2005.01.004. PMID 15806473
- [Background] Perna AF, De Santo NG, Ingrosso D. Adverse effects of hyperhomocysteinemia and their management by folic acid. Miner Electrolyte Metab. 1997;23(3-6):174-8. PMID 9387111
- [Background] Kalantar-Zadeh K, Block G, Humphreys MH, McAllister CJ, Kopple JD. A low, rather than a high, total plasma homocysteine is an indicator of poor outcome in hemodialysis patients. J Am Soc Nephrol. 2004 Feb;15(2):442-53. doi: 10.1097/01.asn.0000107564.60018.51. PMID 14747392
- [Background] Nair AP, Nemirovsky D, Kim M, Geer EB, Farkouh ME, Winston J, Halperin JL, Robbins MJ. Elevated homocysteine levels in patients with end-stage renal disease. Mt Sinai J Med. 2005 Nov;72(6):365-73. PMID 16358160
- [Background] Bayes B, Pastor MC, Bonal J, Junca J, Hernandez JM, Riutort N, Foraster A, Romero R. Homocysteine, C-reactive protein, lipid peroxidation and mortality in haemodialysis patients. Nephrol Dial Transplant. 2003 Jan;18(1):106-12. doi: 10.1093/ndt/18.1.106. PMID 12480967
- [Background] Bowden RG, Wyatt FB, Wilson R, Wilborn C, Gentile M. Homocysteine and vascular access thrombosis in a cohort of end-stage renal disease patients. Ren Fail. 2004 Nov;26(6):709-14. doi: 10.1081/jdi-200037117. PMID 15600264
- [Background] Chen TC, Wang IK, Lee CH, Chang HW, Chiou TT, Lee CT, Fang JT, Wu MS, Hsu KT, Yang CC, Wang PH, Chuang FR. Hyperhomocysteinaemia and vascular access thrombosis among chronic hemodialysis patients in Taiwan: a retrospective study. Int J Clin Pract. 2006 Dec;60(12):1596-9. doi: 10.1111/j.1742-1241.2006.00848.x. Epub 2006 May 16. PMID 16704682
- [Background] Chuang FR, Fang JT, Chen JB, Lin CL, Chen HY, Lee CN, Wang PH, Lee CH. Hyperhomocystinemia and the prevalence of symptomatic atherosclerotic vascular disease in Taiwanese chronic hemodialysis patients: a retrospective study. Ren Fail. 2003 Sep;25(5):765-74. doi: 10.1081/jdi-120024292. PMID 14575285
- [Background] Dennis VW, Robinson K. Homocysteinemia and vascular disease in end-stage renal disease. Kidney Int Suppl. 1996 Dec;57:S11-7. PMID 8941916
- [Background] Suliman ME, Stenvinkel P, Heimburger O, Barany P, Lindholm B, Bergstrom J. Plasma sulfur amino acids in relation to cardiovascular disease, nutritional status, and diabetes mellitus in patients with chronic renal failure at start of dialysis therapy. Am J Kidney Dis. 2002 Sep;40(3):480-8. doi: 10.1053/ajkd.2002.34887. PMID 12200798
- [Background] Bonaa KH, Njolstad I, Ueland PM, Schirmer H, Tverdal A, Steigen T, Wang H, Nordrehaug JE, Arnesen E, Rasmussen K; NORVIT Trial Investigators. Homocysteine lowering and cardiovascular events after acute myocardial infarction. N Engl J Med. 2006 Apr 13;354(15):1578-88. doi: 10.1056/NEJMoa055227. Epub 2006 Mar 12. PMID 16531614
- [Background] Lonn E, Yusuf S, Arnold MJ, Sheridan P, Pogue J, Micks M, McQueen MJ, Probstfield J, Fodor G, Held C, Genest J Jr; Heart Outcomes Prevention Evaluation (HOPE) 2 Investigators. Homocysteine lowering with folic acid and B vitamins in vascular disease. N Engl J Med. 2006 Apr 13;354(15):1567-77. doi: 10.1056/NEJMoa060900. Epub 2006 Mar 12. PMID 16531613
- [Background] Touam M, Zingraff J, Jungers P, Chadefaux-Vekemans B, Drueke T, Massy ZA. Effective correction of hyperhomocysteinemia in hemodialysis patients by intravenous folinic acid and pyridoxine therapy. Kidney Int. 1999 Dec;56(6):2292-6. doi: 10.1046/j.1523-1755.1999.00792.x. PMID 10594808